CLINICAL TRIAL: NCT03041584
Title: Implant-centered Outcomes of Guided Surgery, a 3-year Follow-up: An RCT Comparing Guided Surgery With Non-guided Implant Placement
Brief Title: Dental Implants Placed by Using a Drill Guide Versus Non-guided Placement. Follow-up Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Principal Investigator, Lauren Bernard, Periodontist, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B32220095376
Record Dates: First submitted 2017-01-26; First posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Dental Implant Failure Nos

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Materialise Universal®/ mucosa (Mat Mu) (Experimental)
  Interventions: Procedure: Guided placement; Device: Astra Tech TX implant
- Materialise Universal®/ bone (Mat Bo) (Experimental)
  Interventions: Procedure: Guided placement; Device: Astra Tech TX implant
- FacilitateTM/ mucosa (Fac Mu) (Experimental)
  Interventions: Procedure: Guided placement; Device: Astra Tech TX implant
- FacilitateTM/ bone (Fac Bo) (Experimental)
  Interventions: Procedure: Guided placement; Device: Astra Tech TX implant
- mental navigation (Mental) (Active Comparator)
  Interventions: Procedure: Non-guided placement; Device: Astra Tech TX implant
- pilot-drill template (Templ) (Active Comparator)
  Interventions: Procedure: Non-guided placement; Device: Astra Tech TX implant

INTERVENTIONS:
Procedure: Guided placement — implant placement with use of guide
  Arms: FacilitateTM/ bone (Fac Bo); FacilitateTM/ mucosa (Fac Mu); Materialise Universal®/ bone (Mat Bo); Materialise Universal®/ mucosa (Mat Mu)
Procedure: Non-guided placement — conventional implant placement
  Arms: mental navigation (Mental); pilot-drill template (Templ)
Device: Astra Tech TX implant

SUMMARY:
To assess implant outcomes, both clinical and radiological, in a randomized study on guided implant placement after 3-year follow-up, compared to non-guided treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. An age of at least 18 year
3. Extraction socket healing for at least 6 months

Exclusion Criteria:

1. Unlikely to be able to comply with study procedures
2. History of intravenous bisphosphonate treatment
3. Medical history that makes implant insertion unfavorable
4. Current pregnancy
5. Present alcohol and/or drug abuse
6. Major systemic diseases
7. Untreated, uncontrolled caries and/or periodontal disease
8. History of local irradiation
9. Need for bone grafting and/or sinus lift in the planned implant area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Radiographic outcome | Change between baseline and 3 Year
  Bone loss in mm

SECONDARY OUTCOMES:
probing pocket depth | Change between baseline and 3 Year
  measurement in mm of pocket around implant, 4 per implant
bleeding on probing | Change between baseline and 3 Year
  measurement of presence of bleeding on probing, Yes =1, No=0. 4 per implant
plaque | Change between baseline and 3 Year
  measurement of presence of plaque, Yes =1, No=0. 4 per implant

IPD SHARING:
Plan to Share IPD: Undecided